CLINICAL TRIAL: NCT05709119
Title: Feasibility Study to Investigate the Use of the Oricol™ Sampling Device to Retrieve Vagina Mucus (Wall) Samples for Genomic & Epigenetic Analysis.
Brief Title: Feasibility of the Oricol™ Sampling Device to Retrieve Vagina Mucus (Wall) Samples for Genomic & Epigenetic Analysis.
Acronym: Ellele-01
Status: Completed | Type: Observational
Sponsor: Origin Sciences (Industry)
Collaborators: Royal Infirmary of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: Ellele-01
Record Dates: First submitted 2023-01-24; First posted 2023-02-01 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-01

CONDITIONS: Vagina Disease; Diagnosis
MeSH Terms: conditions — Vaginal Diseases; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — The hydrophilic membrane on the Oricol device allows collection of material from the wall of the vagina including vaginal mucus for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Quantification of human DNA retrieved and DNA fragmentation profile. — The sample will be analysed for material quality and have no impact on the patient's future care.

SUMMARY:
Primary Objective

The primary objective is to explore the feasibility of collecting a vaginal sample using the OriCol™ Sampling Device.

Secondary Objectives

The study has secondary objectives to assess:

1. Acceptability of the sampling technique to both patient and clinician
2. To understand the balloon volume (maximum 80ml) required for effective intra-vaginal sampling.
3. Participant feedback during and after the test for using the OriCol™ Sampling Device using a Visual Analogue Scale
4. Patient discrete choice of Oricol™ versus speculum examination.

DETAILED DESCRIPTION:
The female genital tract is comprised of the vagina, cervix, uterine body, fallopian tubes, and the ovaries. Studies into the dimensions of the vagina have demonstrated there is limited variation, and such variation are not significantly impacted by parity, body size or demographics. The length of the vagina differs depending on measuring techniques and whether the anterior or posterior wall is measured, but on average is between 6 - 10cm in length (OS012-TR001). Vaginal width varies significantly depending on whether this was measured at the level of the introitus, in line with the pelvic floor or more proximally within the tract. Further changes in the vagina are seen in relationship to parity.

As is found in the gastro-intestinal tract, the cervicovaginal tract is, in part, lined with mucus producing goblet cells. The mucus layer also contains shed epithelial cells, microbes and various macromolecules, including antibodies (OS012-TR002). The preliminary results of the colorectal Ori-EGI-02 study, demonstrates that human amplifiable DNA suitable for genomic and epigenetic analysis can be collected from rectal mucus samples (H. N. Humphrey et al. 2022). The rectal mucus samples are collected using the OriCol™ Sampling device, which is inserted into the rectum via a standard proctoscope and then by inflation of a nitrile membrane with 80mL of air.

The current standard examination technique used in gynaecology is a digital vaginal examination (VE) followed by speculum examination. Speculum examination may be performed in the left lateral position (using a Sims Speculum) or in lithotomy (using a Cusco's speculum). Both techniques (and variants) have been in clinical use for over 150 years and allow visual assessment of the vagina and cervix as well as allowing access for diagnostic and/or therapeutic procedures.

The current standard diagnostic investigations for cervical, endometrial, and ovarian malignancy are colposcopy, hysteroscopy, trans-abdominal and trans-vaginal ultrasonography, or CT scanning. Colposcopy requires the insertion of a bivalve speculum into the vagina to directly visualise the cervix. In outpatient hysteroscopy, speculum examination is often carried out to assess the cervix and vagina prior to the procedure. All these investigations take place within a secondary care setting.

The standard Cusco's speculum is bivalved and in the closed state has a length of 80mm and width of 22mm. The volume of the closed lubricated speculum passed into the vagina is 36.3cm3 assuming a closed cylinder. Changes in volume will occur with use. One study assessing the high-pressure zones within the vagina inflated a polyethylene bag of 10cm in length to up to 70cc volume and recorded no adverse effects during the study (OS012-TR001). This suggests that a medical device of 70cc could be inserted into the vagina for diagnostic purposes without discomfort for the patient (Jung et al. 2007)

A review was conducted of the standard Intraspec Contour speculum (Robinson Healthcare Ltd), which is supplied in three sizes: small, medium and large. This was to compare the volume and dimensions of the speculum with the OriCol™ Sampling Device membrane. Origin Sciences Limited have taken measurements of the speculums, as a specification from the manufacturer could not be located.

Due to the characteristics of membrane material of the OriCol™ Sampling Device (PS0025), the height and width of the balloon when inflated to 80ml of air can vary slightly. Inflated membrane quality control (QC) checks during manufacturing indicate that the length of the membrane should not exceed 80mm and the width 63mm. However, the average height of the inflated membrane is approximately 75.2mm and width of 41.3mm. Although the dimensions of the membrane fluctuate slightly between devices, the volume of the inflated membrane stays constant at 65cm3 when inflated with 80mls of air.

The first 40mls of air inserted from the syringe into the membrane push the deflated membrane out of the device. Air inserted above 40mls start to inflate the membrane. This data suggests that at approximate maximum volume (65cm3) the OriCol™ Sampling Device inflated membrane has a smaller volume than a small sized open speculum (~80.9cm3).

There is a current focus on reducing discomfort and increasing compliance in the ability to obtain samples of disease of the female genital tract (Campaign Against Painful Hysteroscopy: Open letter to the UK Department of Health & Social Care (20 October 2022)). Hysteroscopy especially has been the focus on public campaigns to raise awareness of the discomfort associated with this when performed in the Outpatient Setting. Similarly discomfort during sampling of the cervix for pre-malignant change has led to interest in the development of an alternative technology, that is easier to use, has increased patient acceptability and gives a wider range of results leading to greater clinical benefit. As a minimally invasive test, it is important that it's use can be replicated easily, achieve very high levels of compliance, be extremely safe for women and deliver samples that allow high levels of analysis.

In terms of future health economic benefit, the value of the test is the potential reproducibility and ease of use in a variety of clinical settings in primary and secondary care as well as the remote environment.

This feasibility study will address the mechanics of sampling to inform on the technique used in future larger studies.

ELIGIBILITY:
Inclusion Criteria: All participants must meet the following criteria to be eligible for the study:

* Aged 18 years or over
* Able to give voluntary, written informed consent to participate in the study
* Attending a Gynaecology Outpatient Clinic
* Undergoing vaginal speculum examination as part of their routine clinical care

Exclusion Criteria: The following exclusion criteria are applied

* Vaginal, vulval or perineal symptoms make vaginal examination inappropriate.
* Penetrative vaginal sex within the last 24 hours
* Allergy to barrier contraception
* History of allergic reactions to polypropylene and/or nitrile
* Pregnant or suspicion of pregnancy
* Participation in an interventional or pharmaceutical clinical study if treatment/intervention has already commenced
* Previously had a hysterectomy
* Previously had pelvic cancer
* Previously had chemotherapy or pelvic radiotherapy
* Currently undergoing hormone-based treatment for breast or other cancer
* Women with known Hepatitis B, Hepatitis C, HIV or HTLV-II infection, or any other similarly classified human pathogen including prion diseases (Creutzfeldt-Jakob disease).

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — As an intravaginal examination technique, the presence of a natural vagina is required.
Study Population: Patients will be enrolled until 40 samples have been collected and confirmed assessable by the sponsor. Estimated that 45 recruits will be required to collect 40 assessable samples. For this study, 40 Participant samples will be sufficient to fulfil the objectives of the clinical study. The aim is to obtain a variety of samples from pre-, peri- and post-menopausal women to understand if the change in menopausal status affects device acceptability.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
The primary objective is to explore the feasibility of collecting an assessable vaginal sample using the OriCol™ Sampling Device. | Within 3 months of completion of recruitment
  Quantification of human DNA retrieved.

SECONDARY OUTCOMES:
Acceptability of the sampling technique to both patient and clinician | Immediate from test performance
  To assess both ease of use and patient acceptance
To understand the balloon volume (maximum 80ml) required for effective intra-vaginal sampling. | Within 3 months
  Assess variation of vaginal volume and balloon inflation to sample retrieved.
Participant feedback during and after the test for using the OriCol™ Sampling Device using a Visual Analogue Scale | Immediate from test performance
  To assess patient feedback from the test compared to the speculum examination

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Horne, PhD MRCOG, Principal Investigator — Edinburgh Royal Infirmary
Locations (1):
- The Queens Medical Research Institute, Edinburgh, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No